CLINICAL TRIAL: NCT02926898
Title: A Multicenter, 2-Cohort Trial to First Assess the Pharmacokinetic and Safety Profile of a Single Dose of ZX008 (Fenfluramine Hydrochloride) Oral Solution When Added to Standard of Care (Cohort 1), Followed by a Randomized, Double-blind, Placebo-controlled Parallel Group Evaluation of the Efficacy, Safety, and Tolerability of ZX008 as Adjunctive Antiepileptic Therapy to Stiripentol Treatment in Children and Young Adults With Dravet Syndrome (Cohort 2)
Brief Title: A 2-Part Study to Investigate the Dose-Ranging Safety and Pharmacokinetics, Followed by the Efficacy and Safety of ZX008 (Fenfluramine Hydrochloride) Oral Solution as an Adjunctive Therapy in Children ≥ 2 Years Old and Young Adults With Dravet Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX008-1504
Record Dates: First submitted 2016-08-10; First posted 2016-10-06 (Estimated); Results first posted 2022-10-19 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Dravet Syndrome
Keywords: Seizure; Tonic clonic; Epilepsy; Myoclonic; Encephalopathy
MeSH Terms: conditions — Epilepsies, Myoclonic; Seizures; Epilepsy; Brain Diseases | interventions — Fenfluramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 2: ZX008 0.5 mg/kg/day (Experimental): ZX008 0.5 mg/kg/day (maximum 20 mg/day) dose supplied as an oral solution administered twice a day (BID) in equally divided doses with food.
  Interventions: Drug: ZX008 (Fenfluramine Hydrochloride)
- Cohort 2: Matching Placebo (Placebo Comparator): Matching placebo administered twice a day (BID) in equally divided doses with food.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: ZX008 (Fenfluramine Hydrochloride) — ZX008 0.5 mg/kg/day (maximum 20 mg/day). ZX008 drug product is an oral aqueous solution of fenfluramine hydrochloride buffered to pH 5 and provided in concentrations of 2.5 mg/mL.
  *Note: The 0.5 mg/kg/day dose of ZX008 fenfluramine hydrochloride in this study is equivalent to 0.4 mg/kg/day (maximum 17 mg/day) dose of fenfluramine base.
  Arms: Cohort 2: ZX008 0.5 mg/kg/day
Drug: Matching Placebo — Matching Placebo
  Arms: Cohort 2: Matching Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, and efficacy of ZX008 (fenfluramine hydrochloride) when added to adjunctive antiepileptic stiripentol treatment in children and young adults with Dravet syndrome.

DETAILED DESCRIPTION:
This is a multicenter, 2-cohort trial to first assess the pharmacokinetic and safety profile of a single dose of ZX008 (fenfluramine hydrochloride) oral solution when added to a standard Dravet syndrome treatment regimen containing valproate (VPA) and clobazam (CLB), with or without stiripentol (STP) (Cohort 1), followed by a randomized, double-blind, placebo-controlled parallel group evaluation of the efficacy, safety, and tolerability of ZX008 as adjunctive therapy for seizures in children and young adults with Dravet syndrome (Cohort 2).

ELIGIBILITY:
Key Inclusion Criteria:

* Subject must be male or non-pregnant, non-lactating female, aged 2 to 18 years (inclusive).
* Subject must have documented medical history to support a clinical diagnosis of Dravet syndrome, where convulsive seizures are not completely controlled by current antiepileptic drugs.
* Subject must be receiving a therapeutically relevant and stable dose of stiripentol (STP) plus clobazam (CLB) and/or valproate (VPA), and for at least 4 weeks prior to screening and be expected to remain stable throughout the study (Cohort 2 only).
* Subject must be receiving a stable dose of CLB and VPA, administered twice daily (BID), to be eligible for Dose Regimen 1 and 2, or subject must be receiving a stable dose of CLB, VPA, and STP, administered BID, to be eligible for Dose Regimen 3 (Cohort 1 only).

Key Exclusion Criteria:

* Subject has a known hypersensitivity to fenfluramine or any of the excipients in the study medication.
* Subject has pulmonary arterial hypertension.
* Subject has a current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction, or stroke.
* Subject has a current or recent history of anorexia nervosa, bulimia, or depression within the prior year that required medical treatment or psychological treatment for a duration greater than 1 month.
* Subject has a current or past history of glaucoma.
* Subject is receiving concomitant therapy with: centrally acting anorectic agents; monoamine-oxidase inhibitors; any centrally acting compound with clinically appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; triptans, atomoxetine, or other centrally acting noradrenergic agonists; cyproheptadine, and/or cytochrome P450 (CYP) 2D6/3A4/2B6 inhibitors/substrates.
* Subject is currently taking carbamazepine ,oxcarbazepine, eslicarbazepine, phenobarbital, or phenytoin, or has taken any of these within the past 30 days, as maintenance therapy.
* Subject has a positive result on urine tetrahydrocannabinol (THC) panel or whole blood cannabidiol (CBD) at the Screening Visit.
* Subject has a clinically significant condition, or has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to the Screening Visit, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - Children'S Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children'S Hospital of Chicago, Chicago, Illinois
  - Children'S Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
- Canada (2):
  - Bc Children'S Hospital Division of Neurology, Vancouver, British Columbia
  - Chu Sainte-Justine Hospital Neurology Clinic, Montreal, Quebec
- France (9):
  - Chu Amiens Picardie Service de Neurologie Pédiatrique, Amiens
  - Chu de Bordeaux Hôpital Des Enfants, Bordeaux
  - HÔPITAL FEMME-MÈRE-ENFANT Hôpital Service de Neurologie Pédiatrique, Bron
  - Chru de Lille Hôpital Roger Salengro, Lille
  - Hôpital de La Timone, Service de Neuro-Métabolisme Pédiatrique, Marseille
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert-Debré, Paris
  - Chu de Toulouse - Hôpital Des Enfants, Toulouse
  - Hôpital D'Enfants Chur de Nancy, Vandœuvre-lès-Nancy
- Germany (3):
  - Krankenhaus Mara, Epilepsie-Zentrum Bethel, Bielefeld
  - Universitätsklinikum Schleswig-Holstein, Klinik Für Neuropädiatrie, Kiel
  - Kleinwachau Sächsisches Epilepsiezentrum Radeberg, Radeberg
- Netherlands (2):
  - Epilepsiecentrum Kempenhaeghe, Heeze
  - Stichting Epilepsie Instellingen Nederland, Zwolle
- Spain (3):
  - Hospital Sant Joan de Déu Barcelona, Barcelona
  - Hospital Ruber Internacional-Servicio de Neurología, Madrid
  - Cliníca Universidad de Navarra Nidad de Neuropediatría, Pamplona
- United Kingdom (4):
  - Royal Hospital For Children, Queen Elizabeth University, Institute of Neurosciences Hospital, Glasgow, Scotland
  - Alder Hey Children'S Nhs Foundation Trust, Littlewood'S Neurosciences Unit, Liverpool
  - Evelina London Children'S Hospital, Paediatric Neurosciences, London
  - Great Ormond Street Hospital For Children Nhs Foundation Trust, London

REFERENCES:
- [Result] Nabbout R, Mistry A, Zuberi S, Villeneuve N, Gil-Nagel A, Sanchez-Carpintero R, Stephani U, Laux L, Wirrell E, Knupp K, Chiron C, Farfel G, Galer BS, Morrison G, Lock M, Agarwal A, Auvin S; FAiRE, DS Study Group. Fenfluramine for Treatment-Resistant Seizures in Patients With Dravet Syndrome Receiving Stiripentol-Inclusive Regimens: A Randomized Clinical Trial. JAMA Neurol. 2020 Mar 1;77(3):300-308. doi: 10.1001/jamaneurol.2019.4113. PMID 31790543
- [Derived] Cross JH, Galer BS, Gil-Nagel A, Devinsky O, Ceulemans B, Lagae L, Schoonjans AS, Donner E, Wirrell E, Kothare S, Agarwal A, Lock M, Gammaitoni AR. Impact of fenfluramine on the expected SUDEP mortality rates in patients with Dravet syndrome. Seizure. 2021 Dec;93:154-159. doi: 10.1016/j.seizure.2021.10.024. Epub 2021 Nov 2. PMID 34768178
- [Derived] Sullivan J, Perry MS, Wheless JW, Galer B, Gammaitoni A. Fenfluramine responder analyses and numbers needed to treat: Translating epilepsy trial data into clinical practice. Eur J Paediatr Neurol. 2021 Mar;31:10-14. doi: 10.1016/j.ejpn.2021.01.005. Epub 2021 Jan 22. PMID 33540241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 study sites in Canada, France, Germany, the Netherlands, Spain, the United Kingdom, and the United States enrolled participants for Study 1504 Cohort 2.
Pre-assignment Details: A total of 115 subjects were screened for eligibility to participate in Study 1504 Cohort 2. Of these, 87 subjects were enrolled and randomized.
Groups:
- Cohort 2: ZX008 0.5 mg/kg/Day: ZX008 0.5 mg/kg/day (maximum 20 mg/day) administered twice a day (BID) in equally divided doses.
- Cohort 2: Matching Placebo: Matching placebo administered twice a day (BID) in equally divided doses.
Period: Overall Study
Arm/Group | Cohort 2: ZX008 0.5 mg/kg/Day | Cohort 2: Matching Placebo
Started | 43 | 44
Completed | 36 | 41
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: ZX008 0.5 mg/kg/Day: ZX008 0.5 mg/kg/day (maximum 20 mg/day) dose administered twice a day (BID) in equally divided doses.
- Total: Total of all reporting groups
Arm/Group | Cohort 2: ZX008 0.5 mg/kg/Day | Cohort 2: Matching Placebo | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: years]
  Cohort 2 | 8.8 (4.56) | 9.4 (5.05) | 9.1 (4.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Cohort 2: Female | 20 | 17 | 37
  Cohort 2: Male | 23 | 27 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 25 | 22 | 47
  Unknown or Not Reported | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Cohort 2: American Indian or Alaska Native | 0 | 0 | 0
  Cohort 2: Asian | 2 | 1 | 3
  Cohort 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Cohort 2: Black or African American | 1 | 2 | 3
  Cohort 2: White | 23 | 29 | 52
  Cohort 2: More than one race | 0 | 0 | 0
  Cohort 2: Unknown or Not Reported | 17 | 12 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 8 | 2 | 10
  France | 13 | 10 | 23
  Canada | 4 | 3 | 7
  United States | 11 | 11 | 22
  Germany | 0 | 3 | 3
  Spain | 4 | 6 | 10
  United Kingdom | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Convulsive Seizure Frequency (CSF) From the Baseline Period (Baseline) to the Combined Titration + Maintenance (T+M) Period
Description: Monthly (28 day) convulsive seizure frequency (CSF) was based on electronic diary data obtained for each participant. Convulsive seizures included hemiclonic, focal with clear observable motor signs, generalized tonic clonic, secondarily generalized tonic clonic, tonic, clonic, and drop seizures (tonic/atonic). The number of convulsive seizures reported during the entire time interval was divided by the number of nonmissing diary days and the result was then multiplied by 28 to get a 28-day CSF.
Time Frame: 15 weeks (combined Titration + Maintenance Period)
Population: Modified intent-to-treat (mITT) Population, defined as all randomized subjects who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available.
Measure: Mean (Standard Deviation); unit: Convulsive seizures per 28 days
Arm/Group | Cohort 2: ZX008 0.5 mg/kg/Day | Cohort 2: Matching Placebo
Number analyzed (Participants) | 43 | 44
Convulsive seizures per 28 days | -3.18 (44.121) | -0.65 (8.767)
Statistical Analysis 1: Comparison: Cohort 2: ZX008 0.5 mg/kg/Day vs Cohort 2: Matching Placebo; Test type: Superiority; p < 0.001, ANCOVA — Analysis of covariance (ANCOVA) model with treatment group (ZX008 or placebo) and age group (< 6 years, ≥ 6 years) as factors, and with log baseline frequency as a covariate, and log CSF as the outcome variable; Percent difference = -54.0, 95% CI 2-sided [-67.2 to -35.6]

2. Secondary Outcome: Percentage of Participants Who Achieved ≥ a 50% Reduction in Convulsive Seizure Frequency From Baseline to the Combined Titration + Maintenance Period
Description: Percentage of participants who achieved ≥ a 50% reduction in convulsive seizure frequency from Baseline compared to the combined Titration + Maintenance Periods in the ZX008 0.5 mg/kg/day vs placebo groups.
Time Frame: 15 weeks (combined Titration + Maintenance Period)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: ZX008 0.5 mg/kg/Day | Cohort 2: Matching Placebo
Number analyzed (Participants) | 43 | 44
Percentage of participants | 53.5 | 4.5
Statistical Analysis 1: Comparison: Cohort 2: ZX008 0.5 mg/kg/Day vs Cohort 2: Matching Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; A logistic regression model using a categorical response variable as a function of Treatment group, Baseline seizure frequency, and age group

3. Secondary Outcome: Longest Convulsive Seizure-Free Interval (Days)
Description: Comparison of the duration of the longest convulsive seizure-free interval (days) during the combined Titration + Maintenance Periods for the ZX008 0.5 mg/kg/day and placebo groups.
Time Frame: 15 weeks (combined Titration + Maintenance Period)
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 2: ZX008 0.5 mg/kg/Day | Cohort 2: Matching Placebo
Number analyzed (Participants) | 43 | 44
Days | 22.0 [3.0 to 105.0] | 13.0 [1.0 to 40.0]
Statistical Analysis 1: Comparison: Cohort 2: ZX008 0.5 mg/kg/Day vs Cohort 2: Matching Placebo; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The period of observation for Adverse Events extended from the time the subject gave informed consent until the end of the Follow-up Visit (up to Day 120 [Visit 13]).
Arm/Group | Cohort 2: ZX008 0.5 mg/kg/Day | Cohort 2: Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 6/43 | 7/44
Other Adverse Events (participants affected / at risk) | 42/43 | 42/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 2: ZX008 0.5 mg/kg/Day (N=43) | Cohort 2: Matching Placebo (N=44)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 4
Seizure cluster (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 2: ZX008 0.5 mg/kg/Day (N=43) | Cohort 2: Matching Placebo (N=44)
Diarrhea (Gastrointestinal disorders) | 10 | 3
Fatigue (General disorders) | 11 | 2
Pyrexia (General disorders) | 11 | 4
Bronchitis (Infections and infestations) | 5 | 2
Blood glucose decreased (Investigations) | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 19 | 5
Lethargy (Nervous system disorders) | 6 | 2
Seizure (Nervous system disorders) | 2 | 7
Constipation (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 3 | 2
Ear Infection (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 7 | 15
Rhinitis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Blood pressure diastolic increased (Investigations) | 0 | 3
Blood pressure increased (Investigations) | 0 | 3
Echocardiogram abnormal (Investigations) | 4 | 0
Weight decreased (Investigations) | 4 | 1
Generalized tonic-clonic seizure (Nervous system disorders) | 0 | 3
Somnolence (Nervous system disorders) | 3 | 3
Status epilepticus (Nervous system disorders) | 5 | 0
Tremor (Nervous system disorders) | 5 | 0
Abnormal behavior (Psychiatric disorders) | 4 | 1
Irritability (Psychiatric disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT02926898/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT02926898/SAP_001.pdf